CLINICAL TRIAL: NCT05969262
Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites During the Occurrence and Development of Head and Neck Cancer in Southern China
Brief Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites of Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-123
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Metabolite
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head and neck cancer patients: Patients who meet the diagnostic criteria of the Guidelines for Diagnosis and Treatment of Head and Neck Cancer
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- Healthy people: Healthy people without liver related medical history or other diseases known to affect blood lipid/protein metabolism.
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy

INTERVENTIONS:
Diagnostic Test: Proteomics technology and liquid biopsy — using proteomics technology and liquid biopsy to investigate the changes of plasma and urine metabolites in different liver diseases during the development of liver cancer by collecting residual blood and urine from routine diagnosis and treatment or physical examination

SUMMARY:
Dynamic changes in the internal environment of the body are important clues for early detection, diagnosis and even cure of head and neck tumors. This project uses the combination of proteomics technology and liquid biopsy to provide more primary prevention strategies for early intervention, secondary prevention strategies for early detection and treatment, and clues for the study of the mechanism of dynamic evolution of head and neck tumors.

DETAILED DESCRIPTION:
Head and neck cancer is the seventh most common malignant tumor in the world, and China is a country with a high incidence of head and neck cancer. Dynamic changes in the internal environment of the body are important clues for early detection, diagnosis and even cure of head and neck tumors. The occurrence and development of head and neck cancer is complex, so it is particularly important to explore the changes of internal environment in its clinical pathway. Therefore, we conducted this study to investigate the changes of plasma and urine metabolites during the development of head and neck cancer.

(1) Retrospective cohort: 250 patients were recruited, including 125 patients with Head and neck cancer and 125 healthy people.,(2) Prospective cohort: 250 patients were recruited, including 125 head and neck cancer patients and 125 healthy people. During the course of the study, the subjects will not be given or provided with any randomized or any treatment driven by the study protocol. If it is clinically applicable, the treatment physician shall make the treatment decision and choose the treatment plan at his discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Head and neck cancer patients

   * Age 18-75 years old;
   * Male or non-pregnant female;
   * Patients who were normatively diagnosed as head and neck tumors according to the WHO standards of 2017;
   * The general situation is good: KPS score ≥70;
   * No other malignant tumors.
2. Healthy people

   * Age 18-75 years old;
   * Male or non-pregnant female;
   * No history of head and neck related diseases or other diseases known to affect blood lipid/protein metabolism.

Exclusion Criteria:

* Previous history of non-research related head and neck conditions or other known effects on blood metabolism (except for controlled type 2 diabetes);
* With a history of other malignancies (except cell carcinoma and cervical carcinoma in situ);
* Diseases that require long-term use of immunosuppressive drugs (including steroids), including but not limited to congenital or acquired immunodeficiency disorders or active central nervous system rotations, metastatic cancer, active infection, or uncontrolled heart disease;
* Concurrent with other uncontrolled serious medical conditions, such as unstable heart disease that requires treatment Disease, poorly controlled diabetes (fasting blood glucose > 1.5× the upper limit of normal), mental illness and a history of severe allergies.
* BMI less than 18 or greater than 25.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who met the diagnosis and criteria of head and neck cancer and were hospitalized in Southern Hospital of Southern Medical University.Subjects agreed to participate in the study and signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Achieve the expected number of enrolled cases | 3 years
  1. Retrospective cohort: 250 patients were recruited, including 125 patients with head and neck cancer, 125 healthy people.
  2. Prospective cohort: 250 patients were recruited, including 125 head and neck cancer patients and 125 healthy people.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China